CLINICAL TRIAL: NCT06989996
Title: Study of Human Ocular Hemodynamics by Holography Dopple
Acronym: HoLoEye
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P24-02
Record Dates: First submitted 2025-05-02; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Glaucoma; Retinal Vascular Disorder
Keywords: glaucoma; pachychoroid,; carotid stenosis
MeSH Terms: conditions — Glaucoma; Carotid Stenosis

STUDY DESIGN:
Intervention Model Description: * Patients wirhs ocular disease: patients with glaucoma and patients with choroidal disease
  * Participants without ocular disease: healthy volunteers and patients with carotid stenosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Ocular Disease (Experimental): Holodoppler Imaging, Acquisition of useable video images
  Interventions: Device: Images Acquisition
- participants without Ocular Disease (Active Comparator): Holodoppler Imaging, Acquisition of useable video images
  Interventions: Device: Images Acquisition

INTERVENTIONS:
Device: Images Acquisition — Acquisition of useable video images

SUMMARY:
Prospective, interventional, non-randomized, open-label study, multi-center, Gehan-designed study with sequential inclusions in each subgroup, ranging from 4 subjects to a maximum 37 subjects per subgroup included

DETAILED DESCRIPTION:
Retinal perfusion can be affected by a number of local or general pathologies; however, there is currently no commercially available device to provide accurate measurements of retinal blood flow. The company Quantel Medical is developing a medical imaging device HoloDoppler (hereinafter referred to as the "HoloDoppler system"). system. In order to better define its medical utility, we aim to evaluate its reproducibility and accuracy in healthy subjects and those with conditions that may affect ocular blood flow.

ELIGIBILITY:
Inclusion Criteria:

Criteria common to both populations ( patients and healthy volunteers) :

* Age ≥ 18 years and < 75 years;
* Having received informed information about the study and having signed a consent to participate in the study;
* Affiliated or covered by social security

Criteria for healthy volunteers :

No ocular or systemic disease deemed to affect ocular circulation by an investigator

Specific criteria for patients:

* Subjects usually followed at one of the recruiting centers;
* Patients with chronic glaucoma, for whom a therapeutic modification is planned in the short term;
* Patients with carotid stenosis;
* Patients with choroidal pathology: pachychoroidism having led to pigment epithelium anomalies.

Exclusion Criteria:

* For all participants:
* Persons covered by articles L1121-5 to L1121-8 of the CSP (all protected persons: pregnant women, parturients, nursing mothers, persons deprived of their liberty by judicial decision or administrative decision, minors, and persons under legal protection: guardianship or curatorship);
* Women of childbearing age not using an effective method of contraception, or positive pregnancy test (blood or urine);
* Participants allergic to tropicamide when using pupillary dilatation;
* Inability of the subject to maintain a stable sitting position for research procedures;
* Temporary contraindication to HoloDoppler:

  * Patient suffering from viral conjunctivitis or any other infectious disease;
  * Patient with skin lesions on the neck or forehead, for which contact with a chin strap is not recommended.
* Impossibility of making acquisitions of interest (e.g. due to a pupil diameter that is too small, advanced cataracts, nystagmus, etc.).
* Wearing glasses or contact lenses to correct a refractive disorder is not considered a criterion for non-inclusion.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of blood flow monitoring | 15 minutes
  Evaluate the feasibility of retinal blood flow measurement with HoloDoppler imaging
Assessment of the reproducibility of blood flow measurements | 15 minutes
  Determine the reproducibility of retinal blood flow measurements with holodoppler at 15 minutes with the same operator and two different operators
  This is an evaluation of image quality in terms of operation according to the following scheme.
  Quality assessment:
  - Sufficient quality : Yes Or No
  If no, tick yes, below and fill in the cause:
  Insufficient quality: ☒ yes ☐ no
  Cause:
  * Technical problem Or
  * Patient-related problem (inability to fix, or comply with procedure, etc.).
statistical precision measurements by intra-class coefficient (ICC) | 15 minutes
  evaluate the accuracy of measurements or assessments by different operators the HoloDoppler system

CONTACTS AND LOCATIONS:
Overall Officials: Michel PAQUES, Principal Investigator — Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts